CLINICAL TRIAL: NCT06966583
Title: Safety and Preliminary Efficacy Study of NAD+Supplements (NMN) Combined With Radioimmunotherapy in Advanced Non Small Cell Lung Cancer Patients
Brief Title: NAD+ Supplement（NMN）With Radioimmunotherapy in Advanced NSCLC
Acronym: NMN
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, You Lu, Chair of Division of Thoracic Tumor Multimodality Treatment, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HX257253; 257253 (Other Grant/Funding Number: West China Hospital)
Record Dates: First submitted 2025-04-02; First posted 2025-05-12 (Actual); Last update posted 2025-05-12 (Actual); Status verified 2025-05

CONDITIONS: Solid Tumor; Non Small Cell Lung Cancer
Keywords: Radiotherapy; Stereotactic Ablative Radiotherapy; Immunotherapy; NMN
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy; Immunotherapy; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NAD supplement NMN+PD-1 inhibitor+radiotherapy (Experimental): This is a dose escalation study that involves administering radiation therapy (RT) doses, PD-1 inhibitors, and NAD supplements
  Interventions: Dietary Supplement: NAD supplement; Radiation: Radiotherapy; Drug: Immunotherapy

INTERVENTIONS:
Dietary Supplement: NAD supplement — NAD supplement NMN：NMN12000 GeneHarbor
  Other Names: NMN
Radiation: Radiotherapy — Low Dose Radiotherapy or Stereotactic Ablative Radiotherapy or Conventional Radiotherapy
Drug: Immunotherapy — PD-1 inhibitor
  Other Names: PD-1 inhibitor

SUMMARY:
This is a phase I, single center (West China Hospital, Sichuan University) study aimed at investigating the safety and efficacy of NMN supplements combined with chemotherapy and radiation therapy for second-line and above treatment of advanced NSCLC.

DETAILED DESCRIPTION:
This study is a prospective, phase I, dose exploration (NMN dose escalation) clinical trial of radiotherapy combined with immunotherapy for advanced non-small cell carcinoma. The aim is to evaluate the safety and efficacy of NAD supplementation combined with radiotherapy and immunotherapy (+/- chemotherapy) in 20 patients with advanced non-small cell carcinoma who failed first-line treatment.The patient received PD-1 inhibitor combined with radiation therapy for the primary lesion and/or metastatic site (excluding intracranial lesions), and orally took NAD+supplement NMN. Regular monitoring indicators include ORR and PFS of patients' radiation therapy lesions and other observed lesions, medication safety, biomarkers, and OS.

Tolerance observation will be conducted using a 3+3 NMN dose escalation approach until dose limiting toxicity (DLT) is observed in at least 2 out of 3-6 subjects, or tolerance observation of the study treatment will be conducted。 3 cohorts with increasing dose levels:NMN12000 GeneHarbor:150mg,Oral administration, once a day;Second dose group: NMN12000 GeneHarbor:150mg,Oral administration, twice a day;Third dose group: NMN12000 GeneHarbor:150mg,Oral administration,3 times a day.

ELIGIBILITY:
Inclusion Criteria:

1. According to the 8th edition TNM staging of lung cancer by the International Association for the Study of Lung Cancer and the Joint Committee on Cancer Classification in the United States, metastatic (stage IV) non-small cell lung cancer with histological or cytological evidence that cannot be treated surgically and cannot receive curative concurrent chemoradiotherapy, and has received at least first-line treatment.
2. At least 2 measurable target lesions (RECIST v1.1 standard), intracranial lesions are not included as radiation therapy lesions or observation lesions due to immune exemption, liver lesions are not included as observation lesions due to immune exemption, and bone lesions are not included as observation lesions due to non measurability. For a lesion that has previously received radiotherapy, only when there is clear disease progression after radiotherapy can it be considered a target lesion. The patient plans to undergo radiotherapy combined with PD-1 inhibitors, or is currently receiving PD-1 inhibitor treatment and has undergone or plans to undergo radiotherapy within one month from the date of enrollment.
3. Agree to provide tumor tissue specimens, which can be previously archived or freshly obtained, for the detection of biomarkers.
4. Voluntarily sign a written informed consent form. The informed consent form must be signed before any protocol related procedures (which are not part of the subject's routine medical care) are carried out. The subject signs the informed consent form and signs the date. Participants must be willing and able to comply with the scheduled visits, treatment plans, laboratory tests, and other requirements of the study. At the time of signing the informed consent form, both males and females are eligible for age between 18 and 75 years old.
5. The physical fitness score of the Eastern Cooperative Oncology Group (ECOG) in the United States is 0 or 1, with an expected survival period of ≥ 3 months.
6. Can provide confirmation of EGFR through tissue based testing, ALK and ROS1 are both reported as wild-type. For non squamous NSCLC patients who have not been confirmed to have wild-type EGFR and wild-type ALK, tumor samples (archived or fresh, primary or metastatic) need to be collected before enrollment for evaluation of EGFR and ALK testing (in local or central laboratories). If there is no archived tumor tissue, fresh tumor biopsy samples must be collected at baseline.
7. The laboratory test results during the screening period indicate that the subjects have good organ function (no blood components or cell growth factors are allowed to support treatment within the first 2 weeks of randomization): Hematology: i. Absolute neutrophil NEC ≥ 1.5 × 10 ^ 9/L; Ii. Platelet count ≥ 100 × 10 ^ 9/L; Iii. Hemoglobin ≥ 9.0g/dL. B Kidney: i. If the calculated creatinine clearance rate (CrCl) is ≥ 50 mL/min, the Cockcroft Gault formula will be used to calculate CrCl (Cockcroft DW, 1976) CrCL (mL/min)={(140 age) × body weight (kg) × F}/(SCr (mg/dL) × 72), where F=1 for females and F=0.85 for males; SCr=serum creatinine. Liver: i. Serum total bilirubin (TBil) ≤ 1.5 × ULN; For subjects with liver metastasis or confirmed/suspected Gilbert disease, TBil ≤ 3 × ULN ii AST and ALT ≤ 2.5 × ULN; For subjects with liver metastasis, AST and ALT ≤ 5 × ULN d coagulation function: i. International standardized ratio and activated partial thromboplastin time ≤ 1.5 × ULN (unless the subject is receiving anticoagulant therapy and coagulation parameters (PT, INR, and APTT) are within the expected range of anticoagulant therapy at screening).

Exclusion Criteria:

1. Pregnant or lactating women.
2. Researchers believe that any condition that may pose a risk to receiving study treatment or interfere with the evaluation of study treatment, subject safety, or interpretation of study results.
3. Previously received treatment with EGFR antagonists or ALK antagonists.
4. Previously participated in experimental drug studies or received research treatment or used experimental devices within 4 weeks prior to the first administration.
5. Simultaneously enrolled in another clinical study, unless it is an observational, non interventional clinical study or an interventional study with a follow-up period (defined as the time from the first administration to the last administration of the previous clinical study being more than 4 weeks or the study drug having more than 5 half lives).
6. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
7. Suffering from active, known or suspected autoimmune diseases, or having a history of autoimmune diseases, except for vitiligo, hair loss, Graves' disease, psoriasis or eczema that do not require systemic treatment within the past 2 years, hypothyroidism (caused by autoimmune thyroiditis) that only requires stable doses of hormone replacement therapy, and type I that only requires stable doses of insulin replacement therapy, diabetes or childhood asthma that have completely alleviated without any intervention after adulthood, or whose disease will not recur without external triggers.
8. Active or previously recorded inflammatory bowel disease (such as Crohn's disease, ulcerative colitis, or chronic diarrhea).
9. Subjects who require systemic treatment with corticosteroids (>10 mg/day prednisone equivalent dose) or other immunosuppressive drugs within 14 days prior to the first administration. Except for the following: a) If there is no active autoimmune disease, inhaled, ophthalmic, or topical corticosteroids and corticosteroids at doses not exceeding 10mg/day effective dose of prednisone are allowed for treatment. b) The dosage of systemic corticosteroids at physiological doses does not exceed 10 mg/day of prednisone or equivalent doses of other corticosteroids. c) Corticosteroids are used as preventive medication for hypersensitivity reactions (such as medication before CT examination).
10. Known history of primary immunodeficiency virus infection.
11. Suffering from other active malignant tumors within the first 5 years of enrollment. Locally curable cancers (manifested as cured) are excluded, such as basal or cutaneous squamous cell carcinoma, superficial bladder cancer, cervical or breast carcinoma in situ.
12. Having undergone major surgical procedures (defined by the investigator, such as open biopsy, severe trauma, etc.) within 28 days prior to the first administration. Note: For the replacement of intravenous drip tubes, it is acceptable. Within 30 days after the first administration (as determined by the researcher), there are significant surgical plans or complete recovery from previous surgeries. Local surgeries (such as placement of systemic ports, hollow core needle biopsy, and prostate biopsy) are allowed, provided that the surgery is completed at least 24 hours before the first administration of the investigational therapeutic drug.
13. Subjects who have not recovered from the toxicity and/or complications of previous interventions to NCI-CTC AE ≤ 1 degree (excluding hair loss and fatigue) prior to their first medication.
14. History of gastrointestinal perforation and/or fistula within 6 months prior to initial administration.
15. Known history of interstitial lung disease. Exclude subjects highly suspected of having interstitial pneumonia; Or subjects who may interfere with the detection or treatment of suspected drug-related pulmonary toxicity; Or other moderate to severe lung diseases that seriously affect lung function.
16. Known history of active pulmonary tuberculosis (TB). Subjects suspected of having active TB should undergo chest X-ray, sputum examination, and exclusion based on clinical symptoms and signs.
17. Severe infection occurred within 4 weeks prior to the first administration, including but not limited to complications requiring hospitalization, sepsis, or severe pneumonia.
18. Active infections that require systemic treatment.
19. Untreated chronic hepatitis B patients or HBV carriers with chronic hepatitis B virus (HBV) DNA exceeding 500 IU/mL, or active hepatitis C patients should be excluded. Non active HBsAg carriers, treated and stable hepatitis B patients (HBV DNA<500 IU/mL), and cured hepatitis C patients can be enrolled. For HCV antibody positive subjects, they are only eligible to participate in the study if their HCV RNA test results are negative.
20. Individuals who test positive for HIV.
21. Any of the following cardiovascular diseases: a) Evidence of acute or sustained myocardial ischemia; b) Current symptomatic pulmonary embolism; c) Acute myocardial infarction within the first 6 months of randomization; d) Symptomatic congestive heart failure (grade 3 or 4 according to the New York Heart Association functional classification) within the first 6 months of randomization; e) Grade 2 or above ventricular arrhythmia within the first 6 months of randomization; f) Cerebrovascular accident (CVA) or transient ischemic attack within the first 6 months of randomization.
22. Those who have received a live or attenuated vaccine within 30 days prior to the first dose, or those who plan to receive the vaccine during the study period.
23. Known history of severe hypersensitivity reactions to other monoclonal antibodies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events and/or Dose Limiting Toxicities of NMN supplements in RT+ICI treatment | from enrollment through 30 days after last dosing, up to 24 months
  Adverse Events and/or Dose Limiting Toxicity graded per Common Terminology Criteria for Adverse Events (CTCAE) version 5.0

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | up to 24 months after the enrollment
  Investigator assessed PFS according to RECIST v1.1. Progression free survival is defined as time of enrollment to first evidence of progressive disease.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Objective Response Rate (ORR) | up to 24 months after the enrollment
  Investigator assessed ORR using RECIST v1.1 including the all tumor, the tumor undergoing RT and the tumor which do not receive radiotherapy.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Overall Survival (OS) | up to 24 months after the enrollment
  OS is defined as the difference (in months) between the date of study enrollment to the date death due to any cause

OTHER OUTCOMES:
Exploratory indicators | up to 24 months after the enrollment
  The investigators will detect changes in CD4+T absolute count, CD8+T absolute count, CD4+/CD8+T cell ratio, CD38 expression, the concentration of NAD+, granulocyte/lymphocyte ratio, PD-L1 expression, immune related cytokine profile expression levels, etc. in blood/tissue samples by Flow cytometry,ELISA or immunofluorescence experiment.

CONTACTS AND LOCATIONS:
Overall Officials: Jianxin Xue, doctoral, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No
data protection until published

REFERENCES:
- [Background] Wang Y, Wang F, Wang L, Qiu S, Yao Y, Yan C, Xiong X, Chen X, Ji Q, Cao J, Gao G, Li D, Zhang L, Guo Z, Wang R, Wang H, Fan G. NAD+ supplement potentiates tumor-killing function by rescuing defective TUB-mediated NAMPT transcription in tumor-infiltrated T cells. Cell Rep. 2021 Aug 10;36(6):109516. doi: 10.1016/j.celrep.2021.109516. PMID 34380043
- [Background] Song Q, Zhou X, Xu K, Liu S, Zhu X, Yang J. The Safety and Antiaging Effects of Nicotinamide Mononucleotide in Human Clinical Trials: an Update. Adv Nutr. 2023 Nov;14(6):1416-1435. doi: 10.1016/j.advnut.2023.08.008. Epub 2023 Aug 22. PMID 37619764
- [Background] Canner PL, Berge KG, Wenger NK, Stamler J, Friedman L, Prineas RJ, Friedewald W. Fifteen year mortality in Coronary Drug Project patients: long-term benefit with niacin. J Am Coll Cardiol. 1986 Dec;8(6):1245-55. doi: 10.1016/s0735-1097(86)80293-5. PMID 3782631
- [Background] Lv H, Lv G, Chen C, Zong Q, Jiang G, Ye D, Cui X, He Y, Xiang W, Han Q, Tang L, Yang W, Wang H. NAD+ Metabolism Maintains Inducible PD-L1 Expression to Drive Tumor Immune Evasion. Cell Metab. 2021 Jan 5;33(1):110-127.e5. doi: 10.1016/j.cmet.2020.10.021. Epub 2020 Nov 9. PMID 33171124
- [Background] Wu S, Zhang R. CD38-expressing macrophages drive age-related NAD+ decline. Nat Metab. 2020 Nov;2(11):1186-1187. doi: 10.1038/s42255-020-00292-5. No abstract available. PMID 33199923
- [Background] Zhang X, Niedermann G. Abscopal Effects With Hypofractionated Schedules Extending Into the Effector Phase of the Tumor-Specific T-Cell Response. Int J Radiat Oncol Biol Phys. 2018 May 1;101(1):63-73. doi: 10.1016/j.ijrobp.2018.01.094. Epub 2018 Feb 3. PMID 29534901
- [Background] Yin L, Xue J, Li R, Zhou L, Deng L, Chen L, Zhang Y, Li Y, Zhang X, Xiu W, Tong R, Gong Y, Huang M, Xu Y, Zhu J, Yu M, Li M, Lan J, Wang J, Mo X, Wei Y, Niedermann G, Lu Y. Effect of Low-Dose Radiation Therapy on Abscopal Responses to Hypofractionated Radiation Therapy and Anti-PD1 in Mice and Patients With Non-Small Cell Lung Cancer. Int J Radiat Oncol Biol Phys. 2020 Sep 1;108(1):212-224. doi: 10.1016/j.ijrobp.2020.05.002. Epub 2020 May 15. PMID 32417411
- [Background] Park SS, Dong H, Liu X, Harrington SM, Krco CJ, Grams MP, Mansfield AS, Furutani KM, Olivier KR, Kwon ED. PD-1 Restrains Radiotherapy-Induced Abscopal Effect. Cancer Immunol Res. 2015 Jun;3(6):610-9. doi: 10.1158/2326-6066.CIR-14-0138. Epub 2015 Feb 19. PMID 25701325
- [Background] Deng L, Liang H, Burnette B, Beckett M, Darga T, Weichselbaum RR, Fu YX. Irradiation and anti-PD-L1 treatment synergistically promote antitumor immunity in mice. J Clin Invest. 2014 Feb;124(2):687-95. doi: 10.1172/JCI67313. Epub 2014 Jan 2. PMID 24382348
- [Background] Kaur P, Asea A. Radiation-induced effects and the immune system in cancer. Front Oncol. 2012 Dec 17;2:191. doi: 10.3389/fonc.2012.00191. eCollection 2012. PMID 23251903